CLINICAL TRIAL: NCT01335048
Title: Atorvastatin and Clopidogrel HIgh DOse in Stable Patients With Residual High Platelet Activity
Acronym: ACHIDO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ospedale Misericordia e Dolce (Other)
Responsible Party: Principal Investigator, Toso Anna, MD, Ospedale Misericordia e Dolce
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6332011
Record Dates: First submitted 2011-04-11; First posted 2011-04-13 (Estimated); Last update posted 2012-01-26 (Estimated); Status verified 2012-01

CONDITIONS: Stable Angina
Keywords: Clopidogrel; Statins; Platelet reactivity; Point-of-care platelet function test
MeSH Terms: conditions — Angina, Stable | interventions — Atorvastatin; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atorvastatin-Clopidogrel group (Experimental): Patients who receive Atorvastatin 80 mg/day and Clopidogrel 150 mg/day
  Interventions: Drug: atorvastatin and clopidogrel
- Clopidogrel group (Active Comparator): Patients who receive clopidogrel 150 mg daily
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: atorvastatin and clopidogrel — Atorvastatin 80 mg daily + clopidogrel 150 mg daily
  Arms: Atorvastatin-Clopidogrel group
Drug: Clopidogrel — Clopidogrel 150 mg daily
  Arms: Clopidogrel group

SUMMARY:
The purpose of this study is to evaluate if high-dose (80mg/day) atorvastatin might exert an adjunctive anti-platelet effect compared to high-dose clopidogrel (150mg/day) in stable patients with high on-treatment reactivity according to a point-of-care platelet function assay.

DETAILED DESCRIPTION:
This is a prospective, randomized, open-label, control-active trial performed in elective patients candidates to coronary drug eluting stent implantation who presented high-on-treatment platelet reactivity, immediately before coronary intervention (PCI). All patients are treated with aspirin (100 mg/day) and standard-dose clopidogrel (600 mg as loading dose and 75 mg daily as maintenance dose)for at least 7 days before PCI. Platelet function is assessed by the VerifyNow P2Y12 assay (Accumetrics, San Diego, CA). Patients are eligible to be enrolled if they have high-on-treatment reactivity defined as P2Y12 reaction units (PRU) >= 230, immediately before PCI. After PCI, patients are randomized to receive high-dose clopidogrel (150 mg daily) or high-dose atorvastatin (80mg/day) + high-dose clopidogrel (150 mg daily). Study visits and platelet function testing with the VerifyNow P2Y12 test are conducted at 7 and 30 days after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Stable angina
* candidates to drug eluting stent implantation
* High on-treatment platelet reactivity according to a point-of-care platelet function test

Exclusion Criteria:

* chronic therapy with statins
* inability to provide informed consent
* intolerance to statins
* acute or chronic liver failure or ALT > 2 times ULN
* known myopathy
* CKD stage IV or dialysis treatment
* pregnancy or breast-feeding
* malignancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-04; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in on-treatment platelet reactivity at 7 and 30 days | pre-PCI, 7 days and 30 days
  Pharmacodynamic analysis of the randomized groups includes a) assessment of the absolute level of on-treatment reactivity, b) change in on-treatment reactivity, c) rate of high on-treatment reactivity at 7 and 30 days. The platelet reactivity is measured with the VerifyNow P2Y12 test (Accumetrics, SanDiego, CA).

CONTACTS AND LOCATIONS:
Overall Officials: Mario Leoncini, MD, Principal Investigator — Ospedale Misericordia e Dolce, Prato; Anna Toso, MD, Principal Investigator — Ospedale Misericordia e Dolce, Prato
Locations (1):
- Cardiology Department, Ospedale Misericordia e Dolce, Prato, Italy

REFERENCES:
- [Derived] Leoncini M, Toso A, Maioli M, Angiolillo DJ, Giusti B, Marcucci R, Abbate R, Bellandi F. High-dose atorvastatin on the pharmacodynamic effects of double-dose clopidogrel in patients undergoing percutaneous coronary interventions: The ACHIDO (Atorvastatin and Clopidogrel HIgh DOse in stable patients with residual high platelet activity) study. JACC Cardiovasc Interv. 2013 Feb;6(2):169-79. doi: 10.1016/j.jcin.2012.09.013. PMID 23428009